CLINICAL TRIAL: NCT04183595
Title: A Double-blinded, Randomized Controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of N1, N3-bis-(2-Mercaptoethyl) Isophthalamide (NBMI) in the Reduction of Mercury Levels, in Subjects Exposed to Mercury in Colombia
Brief Title: NBMI Treatment in Patients With Mercury Toxicity
Acronym: NBMI-Hg-COL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: EmeraMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Emera008
Record Dates: First submitted 2019-06-19; First posted 2019-12-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Mercury Poisoning
Keywords: Exposure to mercury; NBMI
MeSH Terms: conditions — Mercury Poisoning | interventions — Silicon Dioxide; stearic acid

STUDY DESIGN:
Intervention Model Description: One hundred and sixteen (116) participants will be randomized in a 1:1 ratio, to either one of the two arms of this trial.
  This study will consist of 2 time periods/4 visits
  1. Screening
  2. Day 1 (Treatment start day, 7 days after visit 0)
  3. Day 14 ± 3 days (Treatment end day)
  4. Day 28 ± 3 days (Treatment drug-free follow-up end day)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The research center must assign an unblinded pharmacist or a designated person and a non-blinded CRO monitor, to monitor medication supply and other unblinded documentation of the study.
  Masking through identical capsules and blister in the two arms of intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: NBMI (Study Medication) (Experimental): 600mg / day N1, N3-BIS- (2-MERCAPTOETHYL) ISOPHTHALAMIDE (NBMI) treatment for 14 days, administered as four capsules of 100 mg of NBMI every 24 hours.
  Interventions: Drug: (N1, N3-bis(2- mercaptoethyl)isophthalamide)
- Arm B: Placebo (Placebo Comparator): (Excipients microcrystalline cellulose, silica and magnesium stearate) capsules will be administered every 24 hours for 14 days.
  Interventions: Other: Excipients microcrystalline cellulose, silica and magnesium stearate

INTERVENTIONS:
Drug: (N1, N3-bis(2- mercaptoethyl)isophthalamide) — 600mg / day NBMI treatment for 14 days, administered as four capsules of 100 mg of NBMI every 24 hours, at the start of treatment, the principal investigator or his delegate will verify the intake of the first dose and deliver a blister pack corresponding to the remaining NBMI capsules, at visit day 14 research subjects will be asked to return the packaging with the remaining capsules or not, in order to estimate adherence to treatment.
  Other Names: NBMI
  Arms: Arm A: NBMI (Study Medication)
Other: Excipients microcrystalline cellulose, silica and magnesium stearate — 6 Capsules will be administered every 24 hours for 14 days.
  Other Names: Placebo
  Arms: Arm B: Placebo

SUMMARY:
NBMI (N1, N3-Bis-(2-Mercaptoethyl) Isophthalamide) is a new metal chelator drug proposed as an alternative to the current chelators, and it is widely different; compared to the current chelators, consisting of two cysteamine molecules coupled to a single molecule of dicarboxybenzoate. It is used as a chelating agent and has the designation of an orphan drug, in the EU and USA; in the EU it is used for the treatment of mercury toxicity. It is freely soluble in solutions of dimethylformamide (DMF), dimethyl sulfoxide (DMSO) and sodium hydroxide diluted NaOH, slightly soluble in methanol and acetone, and insoluble in water. Pre-clinical data indicates low to no toxicity, and that it reduces the toxicity associated with acute exposure to Hg2+.

No other chelator has been reported to prevent acute mercury toxicity with only one exposure to the chelator. It has the ability to penetrate cell membranes and cross the blood-brain barrier and chelate Hg2+ in a complex that eliminates the availability of Hg2+ and essentially eliminates toxic effects. The antioxidant properties of NBMI could also reduce the toxicity levels of hydroxyl free radicals immediately, upon entering cells suffering from oxidative stress. It is possible that the combined chelation of Hg2+ and the elimination of hydroxyl free radicals contribute significantly to the protective effects observed with the NBMI.

Previous clinical studies conducted in subjects of the Phase I and Phase II a studies conducted, did not show significant adverse events in patients intoxicated with mercury, all patients who received the study medication have tolerated it well, with only mild or moderate adverse events reported; None of these were considered related to the pharmacological treatment of the study. In addition, there is no potential identified with safety problems in laboratory tests, or vital signs evaluations.

The purpose of this Controlled Single-Center Double-Blind Crossover Clinical Trial Phase II b is to determine the efficacy, safety and tolerability of a 14 day 600mg / day of NBMI (N1, N2-bis-2-mercaptoethyl isophthalamide) Treatment, in the reduction of urinary mercury levels versus placebo, in accidentally exposed subjects to mercury in Colombia.

DETAILED DESCRIPTION:
This is a Controlled Single-Center Double-Blind Crossover Clinical Trial Phase II b conducted in subjects with a history of chronic exposure to mercury in Colombia.

One hundred and sixteen patients (116) will be randomized in a 1:1 ratio, to either one of the two arms of this trial:

Group A:

NBMI (study drug) with an oral dose of 600 mg corresponding to 6 capsules of 100 mg of NBMI every 24 hours for 14 days.

Group B:

Placebo 6 capsules, every 24 hours for 14 days.

This study will consist of 2 time periods/4 visits

1. Screening
2. Day 1 (Treatment start day, 7 days after visit 0)
3. Day 14 ± 3 days (Treatment end day)
4. Day 28 ± 3 days (Treatment drug-free follow-up end day)

After Screening a computer-generated scrambling code will be used for allocation in blocks of 4 to the two treatments. During enrollment, the proportion of subjects with or without a history of previous treatment by chelating will be monitored.

The identity of patients included in the futility analysis will not be provided to the trial team, in order to preserve the blind aspect of the trial.

The trial will be interrupted if the difference between the groups of treatment in the primary assessment is significantly (α = 0.05 unilateral) less than 10% in favor of any of the arms.

A Data Monitoring Committee will be set up to monitor the safety and risk control general benefit. The committee's statistician and epidemiologist will carry out the evaluation.

The identity of the research product associated with each randomization number will be kept hidden for the trial team and for the patients.

The final analysis is planned for when 100% of the patients (116 patients) reach Day 28 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a history of exposure to sources of mercury release by a known event of direct contact with metallic mercury.
* All subjects must have signed and dated an informed consent / assent consent form approved by the IRB in accordance with regulatory and institutional guidelines. This form must be obtained before performing any procedure related to the protocol that is not part of the subject's normal regimen.
* Under age minors must also have a psychological evaluation and documentation of Assent added to the Informed Consent Form.
* Patients with detectable urinary mercury levels >10 ug / L at the time of screening.
* Patients must be willing and able to comply with clinic visits and all study-related procedures.
* Subjects with no previous chelation treatment or who have stopped receiving chelation treatment for more than 3 months will be enrolled.
* Participants must have controlled mercury levels, with no severe clinical manifestations, regardless of what the medical treatment may have been.

Exclusion Criteria:

* A history of known or suspected hypersensitivity or idiosyncratic reactions to the medication or test excipients. Patients with sulfa-drug sensitivity should be excluded from this study.
* Levels of mercury in urine / blood at the time of baseline measurement that are below detection threshold.
* Known history of drug addiction and / or alcoholism.
* Patients with a known medical condition that, in the opinion of the investigator, could increase the risk associated with participation in the study or with the administration of the study medication (s) under blinded conditions or interfere with the interpretation of the security results.
* Patients with major surgery or significant traumatic injury who have not recovered at least 14 days before the first dose of the study medications (s) under blind.
* Subjects with a condition requiring systemic corticosteroid therapy (> 10 mg daily of prednisone equivalent) or other immunosuppressive medications within 14 days before or during treatment are excluded.
* Women with positive pregnancy test (urine sample) at the time of screening; or women who are breastfeeding, or are of childbearing age who disagree with taking contraceptives during treatment and until Day 28 after the last dose.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-05-22 (Estimated); Study Completion 2024-11-22 (Estimated)

PRIMARY OUTCOMES:
Measure the "Change in the subject's urine mercury levels" | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  Evaluation of the difference in mercury levels in the urine as percentage of mercury concentration levels will be determined. The percentage is calculated by comparing baseline mercury concentration levels, against the levels observed at 14-day and 28-days follow-up visits. A rule of three is applied to determine the percentage (%) of change. The analysis of total Hg concentration will be done via Cold Vapor Atomic Absorption spectrometry

SECONDARY OUTCOMES:
Measure the "Change in the subject's blood iron levels" | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  To measure the efficacy, the evaluation of the difference in blood iron levels as the percentages of iron concentration, will be calculated. Immunoturbidimetry Test will be used as an indicator of iron reserves to determine serum ferritin (FS) levels.
Measure the "Change in the subject's blood glucose levels" | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  To measure efficacy, the evaluation of the difference in blood glucose levels, as percentage of glucose concentration, will be determined.
Measure the "Change in the subject's renal function" | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  The difference in scores derived from the CKD-EPI Equation will be evaluated.
Measure the "Frequency and Severity of Adverse Events" | From the first dose of study medication until the Day 56 visit.
  Frequency and Severity of Adverse Events in the 14 day 400mg / day NBMI Treatment Group. Adverse Events will be encoded using the most recent version of the Medical Dictionary for Regulatory Activities.
Measure subject's "Variations in Mental Response ". | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  The European Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) to evaluate quality of life is an instrument to assess the state of health in multiple dimensions. The questionnaire has five questions with Likert (descriptive system) and an analog visual scale (EQ-VAS). The descriptive system defines health in terms of 5 dimensions: mobility, self-care, habitual activities, pain/discomfort and anxiety/Depression. Each dimension has 5 response categories: no problem, mild problems, moderate problems, serious problems and extreme problems. The EQ-VAS marked 0 (worst state of health) -100 (best state of health). The combination of the score in each dimension calculates an index value EQus which is equivalent to the QALY (quality-adjusted life year) value. Thus EQus= 1 is equivalent to QALY = 1, that means a year lived with perfect health, an EQus <1 is equivalent to a year lived with a lower level of health and EQus = 0 is equivalent to being dead.
Measure subject's "Variations in General Clinical examination". | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  A general physical examination of systems and organs will be conducted to determine whether there is or there is not a variation of health status (Yes/No scale). The organs and system that will be examined to determine a general health status are Head and Neck, Oral Cavity, Eyes, Ears, Nose, Cardiovascular System, Chest and Lungs, Abdomen, Skin, Lymphatic System, Neurological System, Renal System, Musculoskeletal System, Appearance).
Measure subject's "Variations in Height". | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  As part of general physical examination variations in participants height will be measured in centimeters comparing measurements in the three visits.
Measure subject's "Variations in Weight". | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  As part of general physical examination variations in participants weight will be measured in kilograms comparing measurements in the three visits.
Mercury intoxication measured by Medical Intoxication Score | Baseline (Before) treatment, Fourteen (14) days after the start of treatment, Fourteen (14) days after the end of treatment
  The medical intoxication score (MIS) is a tool created to identify mercury poisoning in patients. It is a score of ten points that is evaluated by a medical examination, neuromotor tests and an anamnestic questionnaire evaluating 8 elements: 1. Excessive salivation 2. Tremor during work 3. Problems sleeping at night 4. Bluish discoloration of the gums 5. Ataxic gait 6. Dysdiadocokinesia 7. Heel and chin test 8. Proteinuria. Each can have an assigned value of 0 or 1, specific to whether the symptom is absent (0) or present (1) or if the test result is negative (0) or positive (1). The medical score of mercury poisoning is the sum of the values of the elements.
  The worst case of worsening intoxication symptoms would be 10 and a healthy participant will get 0 score. Intoxication will be considered if score is 6 or greater than 6.

OTHER OUTCOMES:
Amalgam | Baseline (Before) treatment
  Presence of amalgam through digital photos
Diet | The patients will keep a food diary during the study (days 1-56).
  During the course of the protocol, all patients will be given a patient's food diary, in which data like type and amount of food intake is self-reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Cadena-Bonfanti, MD, Principal Investigator — Clínica De La Costa Ltda.
Locations (1):
- Clínica de la Costa Ltda., Barranquilla, Atlántico, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordy P, Veiga MM, Salih I, Al-Saadi S, Console S, Garcia O, Mesa LA, Velasquez-Lopez PC, Roeser M. Mercury contamination from artisanal gold mining in Antioquia, Colombia: The world's highest per capita mercury pollution. Sci Total Environ. 2011 Dec 1;410-411:154-60. doi: 10.1016/j.scitotenv.2011.09.006. Epub 2011 Oct 15. PMID 22000915
- [Background] Erkek N, Senel S, Sarac A, Ertan U, Karacan CD. Being alive after a severe inorganic mercury intoxication. Eur J Pediatr. 2010 May;169(5):625-8. doi: 10.1007/s00431-009-1073-2. Epub 2009 Oct 4. PMID 19802724
- [Background] Khan F, Momtaz S, Abdollahi M. The relationship between mercury exposure and epigenetic alterations regarding human health, risk assessment and diagnostic strategies. J Trace Elem Med Biol. 2019 Mar;52:37-47. doi: 10.1016/j.jtemb.2018.11.006. Epub 2018 Nov 14. PMID 30732897
- [Background] Zeitz P, Orr MF, Kaye WE. Public health consequences of mercury spills: Hazardous Substances Emergency Events Surveillance system, 1993-1998. Environ Health Perspect. 2002 Feb;110(2):129-32. doi: 10.1289/ehp.02110129. PMID 11836139
- [Background] Schober SE, Sinks TH, Jones RL, Bolger PM, McDowell M, Osterloh J, Garrett ES, Canady RA, Dillon CF, Sun Y, Joseph CB, Mahaffey KR. Blood mercury levels in US children and women of childbearing age, 1999-2000. JAMA. 2003 Apr 2;289(13):1667-74. doi: 10.1001/jama.289.13.1667. PMID 12672735
- [Background] Park JD, Zheng W. Human exposure and health effects of inorganic and elemental mercury. J Prev Med Public Health. 2012 Nov;45(6):344-52. doi: 10.3961/jpmph.2012.45.6.344. Epub 2012 Nov 29. PMID 23230464
- [Background] Ha E, Basu N, Bose-O'Reilly S, Dorea JG, McSorley E, Sakamoto M, Chan HM. Current progress on understanding the impact of mercury on human health. Environ Res. 2017 Jan;152:419-433. doi: 10.1016/j.envres.2016.06.042. Epub 2016 Jul 18. PMID 27444821
- [Background] Branco V, Caito S, Farina M, Teixeira da Rocha J, Aschner M, Carvalho C. Biomarkers of mercury toxicity: Past, present, and future trends. J Toxicol Environ Health B Crit Rev. 2017;20(3):119-154. doi: 10.1080/10937404.2017.1289834. Epub 2017 Apr 5. PMID 28379072
- [Background] Clarkson TW, Magos L. The toxicology of mercury and its chemical compounds. Crit Rev Toxicol. 2006 Sep;36(8):609-62. doi: 10.1080/10408440600845619. PMID 16973445
- [Background] Clarke D, Buchanan R, Gupta N, Haley B. Amelioration of Acute Mercury Toxicity by a Novel, Non-Toxic Lipid Soluble Chelator N,N'bis-(2-mercaptoethyl)isophthalamide: Effect on Animal Survival, Health, Mercury Excretion and Organ Accumulation. Toxicol Environ Chem. 2012;94(3):616-640. doi: 10.1080/02772248.2012.657199. PMID 22573916
- [Background] Risher JF, Amler SN. Mercury exposure: evaluation and intervention the inappropriate use of chelating agents in the diagnosis and treatment of putative mercury poisoning. Neurotoxicology. 2005 Aug;26(4):691-9. doi: 10.1016/j.neuro.2005.05.004. PMID 16009427
- [Background] George GN, Prince RC, Gailer J, Buttigieg GA, Denton MB, Harris HH, Pickering IJ. Mercury binding to the chelation therapy agents DMSA and DMPS and the rational design of custom chelators for mercury. Chem Res Toxicol. 2004 Aug;17(8):999-1006. doi: 10.1021/tx049904e. PMID 15310232
- [Background] Bose-O'Reilly S, Bernaudat L, Siebert U, Roider G, Nowak D, Drasch G. Signs and symptoms of mercury-exposed gold miners. Int J Occup Med Environ Health. 2017 Mar 30;30(2):249-269. doi: 10.13075/ijomeh.1896.00715. Epub 2017 Mar 22. PMID 28366955
- [Background] Doering S, Bose-O'Reilly S, Berger U. Essential Indicators Identifying Chronic Inorganic Mercury Intoxication: Pooled Analysis across Multiple Cross-Sectional Studies. PLoS One. 2016 Aug 30;11(8):e0160323. doi: 10.1371/journal.pone.0160323. eCollection 2016. PMID 27575533